CLINICAL TRIAL: NCT02808026
Title: A Study to Evaluate Efficacy and Safety of CS-3150 in Japanese Patients With Severe Hypertension (Grade III)
Brief Title: Study of CS-3150 in Patients With Severe Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS3150-A-J304
Record Dates: First submitted 2016-06-17; First posted 2016-06-21 (Estimated); Last update posted 2018-12-21 (Actual); Status verified 2017-03

CONDITIONS: Severe Hypertension
Keywords: severe hypertension; grade III hypertension; mineralocorticoid receptor antagonist
MeSH Terms: conditions — Hypertension | interventions — esaxerenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CS-3150 (Experimental): CS-3150 2.5 to 5mg, orally, once daily after breakfast for 8 weeks
  Interventions: Drug: CS-3150

INTERVENTIONS:
Drug: CS-3150 — CS-3150 2.5 to 5mg, orally, once daily after breakfast

SUMMARY:
To examine antihypertensive effect and safety of administration of CS-3150 in patients with severe hypertension (Grade III).

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged 20 to 80 years at informed consent
* Subjects with severe hypertension, who do not receive any antihypertensive drugs or receive antihypertensive drug (except for potassium-sparing diuretics) during run-in period (Sitting SBP ≥ 180 mmHg or Sitting DBP ≥ 110 mmHg)

Exclusion Criteria:

* Patients who are suspected hypertensive emergency
* Secondary hypertension or malignant hypertension
* Diabetes mellitus with albuminuria
* Serum potassium level < 3.5 or ≥ 5.1 mEq/L (≥ 4.8 mEq/L if receive RA inhibitor)
* eGFR < 60 mL/min/1.73 m^2.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in sitting systolic and diastolic blood pressure | Baseline to end of Week 8

SECONDARY OUTCOMES:
Time course of systolic and diastolic blood pressure | Baseline to end of Week 8
Proportion of patients achieving blood pressure control | Baseline to end of Week 8

CONTACTS AND LOCATIONS:
Locations (1):
- Sapporo, Japan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/